CLINICAL TRIAL: NCT00349583
Title: Efficacy of Topical Cyclosporine Versus Tears for Improving Visual Outcomes Following Multifocal IOL Implantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 1683
Record Dates: First submitted 2006-07-05; First posted 2006-07-07 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-05

CONDITIONS: Cataract; Dry Eye
MeSH Terms: conditions — Cataract; Dry Eye Syndromes | interventions — Cyclosporine

INTERVENTIONS:
Drug: Topical Cyclosporine, Tears

SUMMARY:
The purpose of this study is to evaluate the efficacy on quality of vision and dry eye signs and symptoms in patients undergoing cataract surgery using the ReZoom® multifocal IOL.

ELIGIBILITY:
Inclusion Criteria:

* · Males or females > 50 years old

  * Scheduled to undergo bilateral phacoemulsification with implantation of a multifocal IOL.
  * Likely to complete all study visits and able to provide informed consent
  * Visual potential of 20/25 or better

Exclusion Criteria:

* · Prior use of topical cyclosporine

  * Known contraindications to any study medication or ingredients
  * Active ocular diseases or uncontrolled systemic disease
  * Active ocular allergies

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Eric Donnenfeld, MD, Principal Investigator — Ophthalmic Consultants of Long Island
Locations (1):
- Ophthalmic Consultants of Long Island, Rockville Centre, New York, United States